CLINICAL TRIAL: NCT00325078
Title: Tumor Necrosis Factor Alpha Inhibitor (Lnfliximab, Adalimumab) Treatment for Crohn'S-like Inflammatory Bowel Disease in Chronic Granulomatous Disease: A Phase I/II Study Assessing Clinical and Immune Responses to Treatment and Genetic Influences
Brief Title: Infliximab to Treat Crohn'S-like Inflammatory Bowel Disease in Chronic Granulomatous Disease
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Insufficient patient participation
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 060160; 06-I-0160
Record Dates: First submitted 2006-05-11; First posted 2006-05-12 (Estimated); Results first posted 2015-12-29 (Estimated); Last update posted 2015-12-29 (Estimated); Status verified 2015-11

CONDITIONS: Chronic Granulomatous Disease; Crohn'S-like IBD; Inflammatory Bowel Disease (IBD)
Keywords: Remicade; Crohn's Disease; IBD; CGD Infection; Infliximab; Chorionic Granulomatous Disease; CGD; Inflammatory Bowel Disease
MeSH Terms: conditions — Granulomatous Disease, Chronic; Inflammatory Bowel Diseases; Crohn Disease | interventions — Infliximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Study drug (TNFa inhibitor-infliximab or adalimumab) treated group.
  Interventions: Drug: Infliximab
- Observation (No Intervention): Subjects with IBD without TNFa inhibitor treatment

INTERVENTIONS:
Drug: Infliximab
  Arms: Treatment

SUMMARY:
This study will determine if the drug infliximab is safe for treating inflammatory bowel disease (IBD) in patients with chronic granulomatous disease (CGD). IBD is an inflammation or irritation of the gut that leads to symptoms such as diarrhea, bloating and stomach cramps. CGD is an inherited disease affecting white blood cells called neutrophils in which patients are susceptible to repeated bacterial and fungal infections. They also have a higher incidence of some autoimmune diseases, such as IBD. Infliximab is approved to treat Crohn's disease, an IBD similar to that seen in patients with CGD.

Patients 10 years of age and older with CGD and IBD may be eligible for this study. Candidates are screened with a medical history, physical examination, blood and urine tests, electrocardiogram (EKG), tuberculosis skin test (PPD skin testing), and stool test for the presence of infections. Additional tests may be done, including colonoscopy (procedure using a flexible tube through the rectum to examine the lining of the gut) and imaging studies such as an x-ray, chest CT scan (test using a special x-ray machine), MRI (test using a magnetic field and radio waves), and barium studies (study using a drinkable solution of barium to help enhance the x-ray pictures of the gut).

Participants are divided into patients with IBD symptoms (Group 1) and patients without IBD symptoms (Group 2) for the following procedures:

Group 1

Patients are evaluated every 6 months with a medical history and physical examination for signs and symptoms of IBD. Patients who are taking moderate to high doses of steroid medications have their medication slowly lowered (tapered) and are evaluated every 3 months for a total of 2 years. Patients in this group who start to develop IBD symptoms are moved to Group 2 for treatment with infliximab (see below).

Group 2

Patients in Group 2 receive infliximab infusions at 2-week intervals for three doses. The drug is given over a 2-hour period through a catheter placed in a vein. Patients are evaluated with a medical history, physical exam, and blood tests the day of each dose. One week after the last dose, they have another evaluation, including a colonoscopy. Patients who respond well to infliximab may continue to receive the drug every 2 months for a total of 1 year, with evaluations at every dosing visit. At the end of the first year of receiving infliximab, all patients have follow-up evaluations every 6 months for a total of 2 years.

Group 3

Subjects who volunteer to undergo colonoscopy and research biopsies that serve as controls for evaluation of the patient gut samples.

DETAILED DESCRIPTION:
Chronic Granulomatous Disease (CGD) is an inherited immune disorder involving decreased phagocytic superoxide oxygen radical production, resulting in increased susceptibility to infections. Furthermore, there is a predominance of immune-related inflammatory problems in a subset of CGD patients, such as the inflammatory bowel disease (CGD-IBD). CGD-IBD is often complicated by obstruction, strictures, fissures, fistulae, and extra-intestinal problems. In fact, it is clinically and histologically indistinguishable from Crohn's Disease (CD), another inflammatory bowel disease that affects the general population. Crohn's disease (CD) is a prototypic T helper cell type 1 (Th1) immune disease. Since CGD-IBD bears such close resemblance to CD, it is possible that CGD-IBD is also immune-based. Furthermore, mice studies also support a primarily immune basis for CGD-IBD. However, currently there is little data on this Crohn's-like CGD-IBD in human patients. Treatment for the Crohn's-like CGD-IBD has been primarily oral or topical corticosteroids. Antibiotics have been ineffective and stool cultures typically do not identify clear pathogens. Many patients with the Crohn's-like CGD-IBD disease remain steroid-dependent, thus new therapeutic regimens are needed.

This is a Phase I/II study that will evaluate the safety and efficacy of Tumor Necrosis Factor Alpha Inhibitor (Infliximab or Adalimumab) in CGD patients with symptomatic Crohn's-like IBD. Infliximab and Adalimumab are standard-of-care treatments for moderate to severe CD, with extensive experience using these agents being well documented in terms of safety and efficacy. Preliminary reports from ongoing studies of CD at NIH are encouraging in inducing remission. We will also evaluate changes in immunophenotype and cytokine profiles of peripheral blood and colonic lamina propria lymphocytes following treatment. In addition, we will evaluate the immunophenotype and cytokine profile of blood and mucosal cells in CGD patients, with or without IBD, to determine the CGD-specific cytokine profile. Specific cytokine profiles have been observed in different genetic immunodeficiencies, despite similar IBD clinical manifestation.

Documentation of clinical status will be performed using the Crohn's Disease Activity Index (CDAI). Potential effects of genetic variation (including CGD mutation type) on the expression of IBD in patients with CGD, and their responses to treatment will also be assessed. The long-term goal of this study is to establish better or alternative treatment modalities with low risk profiles for CGD patients with Crohn's-like IBD.

ELIGIBILITY:
* INCLUSION CRITERIA:

Group One

* Must have a confirmed CGD diagnosis
* Must have IBD documented by medical history or documented IBD endoscopically.
* Must not be pregnant or breastfeeding
* Must have a home physician
* Must be willing to submit samples for storage.

Group Two:

* Must have a confirmed CGD diagnosis
* Must have IBD documented by medical history or documented IBD endoscopically.
* Must be symptomatic
* Must have negative results on stool examination for culture of enteric pathogens, such as Salmonella, Shigella, Yersinia, Campylobacter, E. coli O157/H7, Clostridium difficile toxin assay, enteric parasites and their ova such as Cryptosporidia, Cyclospora, Microsporidia and Giardia (by stool enzyme immunoassay [EIA]) prior to the start of receiving TNF? inhibitors.
* Must not be pregnant or breastfeeding
* If of childbearing potential, one must agree to consistently use contraception, while on the study medication.
* Must have a recent chest CT (within 3 months) to confirm absence of tuberculosis (TB) infection
* Must have a home physician
* Must be willing to submit samples for storage.

Group Three:

* Must be willing to undergo upper and lower endoscopy and mucosal biopsies for research purpose
* Must be greater than or equal to 18 years old and weigh greater than or equal to 15 kg.
* Must not be pregnant
* Must be willing to submit samples for storage.

EXCLUSION CRITERIA:

Group One:

- Any condition that, in the investigator's opinion, places the patient at undue risk by participating in the study.

Group Two:

* Any condition that, in the investigator's opinion, places the patient at undue risk by participating in the study
* Positive TB diagnosis
* Patients who are in the at-risk group for treatment such as history of tuberculosis, congestive cardiac failure or myocardial infarction within the last 12 months unstable angina, thrombocytopenia (platelet < 100, 000), uncontrolled hypertension
* Acute systemic or intestinal infection(s)
* Evidence of Hepatitis B or C infection
* Signs and symptoms of hepatotoxicity
* Pregnant or breastfeeding
* History of cancer within the last 10 years
* The presence of certain types of acquired abnormalities of immunity such as HIV, cytotoxic chemotherapy for malignancy could be grounds for possible exclusion if, in the opinion of the investigator, the presence of such disease process interferes with evaluation of a co-existing abnormality of immunity that is a subject of study under this protocol.
* Co-existing Th2-type inflammatory disease
* Current active bowel obstruction, intestinal perforation, or significant GI hemorrhage.
* Live vaccine within 4 weeks prior to therapy or potential need for a live vaccine during the study.
* Unwillingness to undergo testing or procedures associated with this protocol.

Group Three:

* Acute systemic or intestinal infection requiring antibiotics
* Any condition that, in the investigator's opinion, places the patient at undue risk by participating in the study
* The presence of certain types of acquired abnormalities of immunity such as HIV, cytotoxic chemotherapy for malignancy could be grounds for possible exclusion if, in the opinion of the investigator, the presence of such disease process interferes with evaluation of a co-existing abnormality of immunity that is a subject of study under this protocol.
* Unwillingness to undergo testing or procedures associated with this protocol.

Min Age: 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suk S De Ravin, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Vignais PV. The superoxide-generating NADPH oxidase: structural aspects and activation mechanism. Cell Mol Life Sci. 2002 Sep;59(9):1428-59. doi: 10.1007/s00018-002-8520-9. PMID 12440767
- [Background] Segal BH, Leto TL, Gallin JI, Malech HL, Holland SM. Genetic, biochemical, and clinical features of chronic granulomatous disease. Medicine (Baltimore). 2000 May;79(3):170-200. doi: 10.1097/00005792-200005000-00004. PMID 10844936
- [Background] Winkelstein JA, Marino MC, Johnston RB Jr, Boyle J, Curnutte J, Gallin JI, Malech HL, Holland SM, Ochs H, Quie P, Buckley RH, Foster CB, Chanock SJ, Dickler H. Chronic granulomatous disease. Report on a national registry of 368 patients. Medicine (Baltimore). 2000 May;79(3):155-69. doi: 10.1097/00005792-200005000-00003. PMID 10844935
- [Background] Buckner CM, Moir S, Kardava L, Ho J, Santich BH, Kim LJ, Funk EK, Nelson AK, Winckler B, Chairez CL, Theobald-Whiting NL, Anaya-O'Brien S, Alimchandani M, Quezado MM, Yao MD, Kovacs JA, Chun TW, Fauci AS, Malech HL, De Ravin SS. CXCR4/IgG-expressing plasma cells are associated with human gastrointestinal tissue inflammation. J Allergy Clin Immunol. 2014 Jun;133(6):1676-85.e5. doi: 10.1016/j.jaci.2013.10.050. Epub 2013 Dec 25. PMID 24373354

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group: This group comprises patients with Chronic granulomatous disease (CGD) complicated by significant inflammatory bowel disease (IBD). The subjects are treated with a TNFa inhibitor at standard recommended doses for treatment of Crohn's disease. Infliximab is administered as intravenous infusions at 5mg/kg on weeks 0, 2 and 6 for induction and every 6-8 weeks at 5-10mg/kg for maintenance. Adalimumab is administered at 160mg, 60mg, 40mg, 40mg on weeks 0, 2, 4 and 6 via subcutaneous injection.
  Endoscopies and gastrointestinal mucosal biopsies are obtained before treatment, following induction, and again at completion of treatment.
- Observation Group: CGD patients with IBD who are not treated with any study medication and are monitored for rate of infections.
- Control Volunteer: Subjects who volunteer to participate in endoscopy and GI mucosal biopsies to provide controls for the study. The subjects in this arm may be healthy subjects, CGD subjects without GI symptoms, or subjects with Crohn's disease (CD). The rate of infections in the CGD patients without IBD are monitored.
Period: Overall Study
Arm/Group | Treatment Group | Observation Group | Control Volunteer
Started | 8 | 7 | 25
Completed | 3 | 2 | 23
Not Completed | 5 | 5 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group | Observation Group | Control Volunteer | Total
Number analyzed (Participants) | 8 | 7 | 25 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 3 | 0 | 4
  Between 18 and 65 years | 7 | 4 | 25 | 36
  >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 6 | 7
  Male | 7 | 7 | 19 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 2 | 3
  Not Hispanic or Latino | 8 | 6 | 22 | 36
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 6 | 6
  White | 8 | 6 | 15 | 29
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Safety of Study Drug
Description: Number of Infections from Baseline to 1 year
Time Frame: Baseline to 1 year
Population: The volunteer group includes patients with chronic granulomatous disease as well as healthy normal volunteers as controls. Infection rates only pertain to and are counted in subjects with underlying immunodeficiency (chronic granulomatous disease).
Measure: Number; unit: infections
Groups:
- Treatment: This group comprises patients with Chronic granulomatous disease (CGD) complicated by significant inflammatory bowel disease (IBD). The subjects are treated with a TNFa inhibitor at standard recommended doses for treatment of Crohn's disease. Infliximab is administered as intravenous infusions at 5mg/kg on weeks 0, 2 and 6 for induction and every 6-8 weeks at 5-10mg/kg for maintenance. Adalimumab is administered at 160mg, 60mg, 40mg, 40mg on weeks 0, 2, 4 and 6 via subcutaneous injection.
  Endoscopies and gastrointestinal mucosal biopsies are obtained before treatment, following induction, and again at completion of treatment.
- Control Volunteers: Subjects who volunteer to participate in endoscopy and GI mucosal biopsies to provide controls for the study. The subjects in this arm may be healthy subjects, CGD subjects without GI symptoms, or subjects with Crohn's disease (CD). The rate of infections in the CGD patients without IBD are monitored.
Arm/Group | Treatment | Observation | Control Volunteers
Number analyzed (Participants) | 8 | 7 | 8
infections | 5 | 4 | 13

2. Primary Outcome: Efficacy of Treatment With Study Drug
Description: Measured participant Crohn's disease Activity Index (CDAI) values. The CDAI is a tool comprised of clinical and laboratory factors such as stool frequency, consistency, abdominal pain, general well being, weight and blood profile as an objective measure of disease activity. A higher score corresponds to greater severity of inflammatory bowel disease; severe disease conventionally defined as >450, a remission as <150, and a response to treatment as a fall of CDAI of >70 points. Infections and IBD are not expected in healthy control subjects. The greater the score, the more severe the disease, and a score of less than 5 represents clinical remission.
Time Frame: Baseline, 1 year
Population: All participants in the Treatment and Observation Arms with collected CDAI data. The CDAI, a tool validated for Crohn's disease is not applicable to healthy donors or CGD patients without IBD, and therefore not measured in the Control participants.
Measure: Number; unit: Crohn's disease activity Index
Groups:
- Observation: CGD patients with IBD who are not treated with any study medication and are monitored for rate of infections.
Arm/Group | Treatment | Observation
Number analyzed (Participants) | 5 | 5
Crohn's disease activity Index
  CDAI Value #1 at Baseline | 114.4 | 17.5
  CDAI Value #2 at Baseline | 191 | 22.5
  CDAI Value #3 at Baseline | 329.8 | 53
  CDAI Value #4 at Baseline | 505.2 | 159
  CDAI Value #5 at Baseline | 516 | 266.7
  CDAI Value #1 at 1 year | 95.5 | NA — Only patients who completed the year of study drug treatment got a repeat CDAI
  CDAI Value #2 at 1 year | 138 | NA — Only patients who completed the year of study drug treatment got a repeat CDAI
  CDAI Value #3 at 1 year | 185.4 | NA — Only patients who completed the year of study drug treatment got a repeat CDAI
  CDAI Value #4 at 1 year | 259.2 | NA — Only patients who completed the year of study drug treatment got a repeat CDAI
  CDAI Value #5 at 1 year | 295.2 | NA — Only patients who completed the year of study drug treatment got a repeat CDAI

3. Other Pre Specified Outcome: Gut Immune Cell Types and Their Cytokine Profile
Description: Gut Immune cell types and their cytokine profile
Time Frame: 1 year
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: The adverse events reported only relate to events occurring following study drug (TNFa inhibitors) treatment. Group 3 subjects who volunteered for endoscopy/gut biopsies are terminated at completion of the procedure. Baseline infections in endoscopy volunteers are not reported as adverse events.
Arm/Group | Treatment Group | Observation Group | Control Volunteer
Serious Adverse Events (participants affected / at risk) | 2/8 | 0/7 | 0/25
Other Adverse Events (participants affected / at risk) | 3/8 | 1/7 | 0/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=8) | Observation Group (N=7) | Control Volunteer (N=25)
lung infection (Infections and infestations) | 1 | 0 | 0
Nervous system disorders - drug overdose (Nervous system disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group (N=8) | Observation Group (N=7) | Control Volunteer (N=25)
diarrhea (clostridium diff) (Gastrointestinal disorders) | 1 | 0 | 0
Infusion related reaction (General disorders) | 2 | 0 | 0
Infections and infestations, IV line infection (Surgical and medical procedures) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Due to limited subject participation and lack of sustained clinical benefits (1 year), there is insufficient complete data to generate meaningful statistics for the outcome measures. Instead, this data are reported as a case series.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes